CLINICAL TRIAL: NCT00093951
Title: A Multicenter, Randomized, Double-Blind, Placebo-Controlled, Phase II Study of the Efficacy and Safety of SGS742 in Subjects With Mild to Moderate Alzheimer's Disease
Brief Title: SGS742 in Patients With Mild to Moderate Alzheimer's Disease (AD)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Saegis Pharmaceuticals (Industry)
Organization: National Institute on Aging (NIA) (NIH)
Allocation: Randomized | Masking: Double | Purpose: Treatment
Other Study IDs: IA0061
Record Dates: First submitted 2004-10-07; First posted 2004-10-08 (Estimated); Last update posted 2009-12-11 (Estimated); Status verified 2009-02

CONDITIONS: Alzheimer's Disease
Keywords: Alzheimer disease; memory; cognition; GABA(B)receptor antagonist
MeSH Terms: conditions — Alzheimer Disease | interventions — (3-aminopropyl)(n-butyl)phosphinic acid

INTERVENTIONS:
Drug: SGS742

SUMMARY:
The purpose of this trial is to determine the effect of a new drug, SGS742, on memory and cognition in patients with mild to moderate Alzheimer's disease.

DETAILED DESCRIPTION:
SGS742 is a GABA(B) receptor antagonist. It is an orally active drug and possesses neurochemical and psychopharmacologic features that suggest it could improve memory and cognition in humans. The primary objective of the SGS742 clinical trial will be to determine the effect of SGS742 on memory and cognition in individuals diagnosed with mild to moderate Alzheimer's disease. The duration of the study is 3 months with 5 clinic visits.

ELIGIBILITY:
Inclusion Criteria:

* 55 to 90 years of age
* Diagnosed with mild to moderate Alzheimer's disease
* Willing caregiver
* In general good health

Exclusion Criteria:

* Call 1-877-MY-MEMORY and ask to be referred to a study center located near you for entry criteria information.

Prohibited Meds:

* Alzheimer's medications (Aricept, Exelon, Remydl, Nemenda)

Ages: 55 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 280
Dates: Start 2004-04; Primary Completion 2007-09 (Actual); Study Completion 2007-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (58):
- United States (58):
  - Phoenix, Arizona
  - Dedicated Clinical Research, Sun City, Arizona
  - Northwest NeuroSpecialists, PLLC, Tucson, Arizona
  - Clinical Trials Incorporated, Little Rock, Arkansas
  - Margolin Brain Institute, Fresno, California
  - NervePro Research, Irvine, California
  - Center for Neurologic Studies, La Jolla, California
  - Neuro Therapeutics, Inc., Pasadena, California
  - Pacific Research Network, Inc., San Diego, California
  - Affiliated Research Institute, San Diego, California
  - San Francisco Clinical Research Center, San Francisco, California
  - Southern California Clinical Research, Inc., San Marino, California
  - The Mile High Research Center, Denver, Colorado
  - Research Center for Clinical Studies, Inc., Darien, Connecticut
  - Stamford, Connecticut
  - Baumel-Eisner Neuromedical Institute, Inc., Boca Raton, Florida
  - Bradenton Neurology, Inc., Bradenton, Florida
  - Brain Matters, Inc., Delray Beach, Florida
  - Baumel-Eisner Neuromedical Institute, Fort Lauderdale, Florida
  - Berma Research Group, Hialeah, Florida
  - Allied Clinical Trials, The Neurology Group, Miami, Florida
  - Tukoi Institute for Clinical Research, Miami, Florida
  - Baumel-Eisner Neuromedical Institute, Miami Beach, Florida
  - Ocala Neurodiagnostic Center, Ocala, Florida
  - Orange City, Florida
  - Palm Springs, Florida
  - Pompano Beach, Florida
  - Tampa, Florida
  - CSI Research, Decatur, Georgia
  - DeKalb Neurology Associates, LLC, Decatur, Georgia
  - MidAmerica Neuroscience Institute, Lenexa, Kansas
  - Neurology Department, LSU Health Sciences Center, Shreveport, Louisiana
  - Baystate Medical Center, Springfield, Massachusetts
  - SW Medical Associates, Las Vegas, Nevada
  - Paterson, New Jersey
  - Psychopharmacology Research Association of Princeton, P.C., Princeton, New Jersey
  - United Health Services Office of Clinical Trials, Johnson City, New York
  - New York, New York
  - Raleigh Neurology, Raleigh, North Carolina
  - Raleigh, North Carolina
  - Winston-Salem, North Carolina
  - MetroHealth Medical Center, Cleveland, Ohio
  - University Memory and Aging Center, Cleveland, Ohio
  - Toledo, Ohio
  - Lynn Health Science Institute, Oklahoma City, Oklahoma
  - Oregon Center for Clinical Investigations, Inc., Eugene, Oregon
  - Medford, Oregon
  - Bala-Cynwyd, Pennsylvania
  - The Clinical Trial Center, LLC, Jenkintown, Pennsylvania
  - RI Mood & Memory Research Institute, East Providence, Rhode Island
  - Madison, Tennessee
  - Senior Adults Specialty Research, Inc., Austin, Texas
  - Claghorn-Lesem Research Clinic, Ltd., Bellaire, Texas
  - Radiant Research San Antonio, San Antonio, Texas
  - Texas Medical Research Associates, LLC, San Antonio, Texas
  - Grayline Clinical Drug Trials, Wichita Falls, Texas
  - Bennington, Vermont
  - National Clinical Research, Inc., Richmond, Virginia

REFERENCES:
- [Background] Froestl W, Gallagher M, Jenkins H, Madrid A, Melcher T, Teichman S, Mondadori CG, Pearlman R. SGS742: the first GABA(B) receptor antagonist in clinical trials. Biochem Pharmacol. 2004 Oct 15;68(8):1479-87. doi: 10.1016/j.bcp.2004.07.030. PMID 15451390